CLINICAL TRIAL: NCT05870436
Title: A Study on the Diagnostic Value of the Methacholine Choline Provocation Test in the Asthmatic Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: jingping Zheng (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, jingping Zheng, Chief Physician, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: SX20221101
Record Dates: First submitted 2023-05-11; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: asthma diagnosis; Methacholine Choline Provocation Test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive group: The group that conducted the Methacholine Choline Provocation Test with Positive result
  Interventions: Diagnostic Test: Methacholine Choline Provocation Test
- Negative group: The group that conducted the Methacholine Choline Provocation Test with negative result
  Interventions: Diagnostic Test: Methacholine Choline Provocation Test

INTERVENTIONS:
Diagnostic Test: Methacholine Choline Provocation Test — Perform methacholine choline provocation test according to the protocol

SUMMARY:
This study was a multicenter, open, observational study and was divided into two stages; Stage I study includes patients with suspected asthma to observe the diagnostic value and safety of Methacholine Choline Provocation Test. All patients clinically evaluated for bronchial provocation testing were included in the stage II study to further validate the diagnostic value and cutoff value of the methacholine choline provocation test.

DETAILED DESCRIPTION:
This study was a multicenter, open, observational study. The study was divided into two stages; the first stage of the study included a population with suspected asthma and performed a bronchial provocation test, and cumulative provocation dose when forced expiratory volume in one second (FEV1) fell by 20% (PD20 ) data were recorded. Subjects with positive excitation were treated as asthma for 3 months and treatment was considered effective to confirm the diagnosis of asthma. Sensitivity, specificity, and reliability of the methacholine choline provocation test were calculated, and cutoff values were obtained by exploratory analysis based on PD20 values. All patients clinically evaluated for bronchial provocation testing were included in the stage II study to further validate the diagnostic value and cutoff value of the methacholine choline provocation test.

ELIGIBILITY:
Inclusion Criteria:

Stage I study:

* clinically evaluated as suspected asthma but have not been previously diagnosed as asthma and require a bronchial provocation test
* Basal lung function FEV1 ≥ 60%
* Meet the requirements for conducting bronchial excitation tests and pulmonary ventilation examinations
* Not currently suffering from or accompanied by other respiratory diseases, including allergic rhinitis, chronic obstructive pulmonary disease, chronic bronchitis, etc.

Stage II study:

* Basal lung function FEV1 ≥ 60%
* Meet the requirements for conducting bronchial excitation tests and pulmonary ventilation examinations

Exclusion Criteria:

* Have had a fatal asthma attack, or have required mechanical ventilation for an asthma attack within the last 3 months
* Definite hypersensitivity reaction to inhaled stimulants or salbutamol or unexplained urticaria
* Severe impairment of basal pulmonary ventilation (FEV1 < 60% of expected value %, or < 1 L in adults)
* Poor cooperation with basal pulmonary function tests that do not meet quality control requirements
* Other conditions that make a bronchial provocation test or pulmonary ventilation function test inappropriate (e.g., recent presence of severe cardiovascular disease, seizures, uncontrolled hypertension, etc.)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stage I study: patients with one or more symptoms such as wheezing, shortness of breath, cough and chest tightness, clinically evaluated as suspected asthma but not previously diagnosed as asthma and requiring bronchial provocation test, such as patients with suspected asthma without obstructive pulmonary function changes, patients with suspected cough variant asthma (CVA) in chronic cough, patients with recurrent chest tightness episodes suspected of chest tightness variant asthma (CTVA), etc.
  Stage II study: bronchial provocation test is required after clinical evaluation, including patients with suspected asthma, asthma, allergic rhinitis, chronic obstructive pulmonary disease, and chronic bronchitis.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity | Baseline up to 3 months
  The sensitivity, specificity of the test were calculated by the results of the test and whether the patient was finally diagnosed with asthma by performing the methacholine choline provocation test in patients suspected of having asthma

SECONDARY OUTCOMES:
The incidence, severity of adverse events | Baseline up to 1 week
  Safety

OTHER OUTCOMES:
PD20 cutoff value | through study completion, an average of 2 year
  PD20 cutoff values for asthma diagnosis by methacholine choline provocation test

CONTACTS AND LOCATIONS:
Overall Officials: yi Gao, PhD, Principal Investigator — The First Hospital of Guangzhou Medical University
Locations (6):
- China (6):
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Songshan General Hospital, Chongqing, Chongqing Municipality
  - The First Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Tongji Hospital，Tongji Medical College of Hust, Wuhan, Hubei
  - West China Hospital of Sichuan University, Chengdu, Sichaun

IPD SHARING:
Plan to Share IPD: No